CLINICAL TRIAL: NCT07398664
Title: Recombinant Human Adenovirus 5 (H101) Combined With Transcatheter Arterial Chemoembolization (TACE) for the Treatment of Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma: A Single-Center, Prospective Study
Brief Title: H101 Plus TACE for r/m HNSCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Hai Tao, M.D, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCH2025-ONCO-1179
Record Dates: First submitted 2026-01-31; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Oncolytic Virus; TACE
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- H101+TACE (Experimental)
  Interventions: Drug: H101; Procedure: TACE

INTERVENTIONS:
Drug: H101 — H101 combined with transarterial chemoembolization (TACE) for the treatment of recurrent or metastatic head and neck squamous cell carcinoma (r/m HNSCC)
Procedure: TACE — H101 combined with transarterial chemoembolization (TACE) for the treatment of recurrent or metastatic head and neck squamous cell carcinoma (r/m HNSCC)

SUMMARY:
This study evaluates H101 combined with transarterial chemoembolization (TACE) to enhance local tumor killing and immune activation while minimizing toxicity in r/m HNSCC patients.

DETAILED DESCRIPTION:
Recurrent or metastatic head and neck squamous cell carcinoma (r/m HNSCC) carries a dismal prognosis (median OS 7-9 months) and lacks effective treatments. H101, an oncolytic adenovirus approved for nasopharyngeal carcinoma, selectively lyses p53-deficient tumor cells [3]. This study evaluates H101 combined with transarterial chemoembolization (TACE) to enhance local tumor killing and immune activation while minimizing toxicity. Supported by prior safety and efficacy data of both modalities, this regimen represents a promising novel approach for r/m HNSCC.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and under 80 years old.
2. Pathologically confirmed head and neck malignancies (including nasopharyngeal carcinoma, oral cavity cancer, oropharyngeal cancer, laryngeal cancer, hypopharyngeal cancer, salivary gland cancer, nasal cavity and paranasal sinus cancer, etc.); patients who have failed at least two lines of standard treatment (including cetuximab and immuno check point inhibitors).
3. Expected survival ≥3 months.
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0-2.
5. Pre-treatment peripheral blood tests meet the following conditions: neutrophil count >2000/mm³, platelet count >100,000/mm³.
6. Pre-treatment liver and kidney function meet the following: bilirubin <1.5 mg/dL, AST or ALT <1.5 times the upper limit of normal, serum creatinine <1.5 mg/dL, creatinine clearance >60 mL/min.
7. Agreement to follow the trial treatment plan and visit schedule, voluntary participation, and written informed consent.

Exclusion Criteria:

1. Expected survival less than 3 months.
2. Positive pregnancy test for women of childbearing age.
3. Concurrent diseases or conditions that affect the patient's ability to enroll normally or safety during the study period.
4. Active psychiatric disorders or other psychological conditions that affect the patient's ability to sign the informed consent or understand the study.
5. Severe coagulation abnormalities and/or active infection requiring intravenous anti-infective therapy.
6. History of another malignancy within 5 years prior to screening, except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or microscopic papillary thyroid carcinoma that have been treated with potential curative therapy.
7. Severe cardiac arrhythmia or conduction abnormalities, and clinically uncontrolled hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >90 mmHg).
8. Adverse reactions from prior anti-tumor treatments have not recovered to CTCAE version 5.0 Grade <1 (except for toxicities judged by the investigator to pose no safety risk, such as alopecia, Grade 2 peripheral neuropathy, etc.).
9. History of infectious diseases, such as positive HIV antibody test, active hepatitis B (defined as HBsAg positive during screening, with HBV-DNA levels above the upper limit of normal at the local laboratory), or hepatitis C (defined as positive HCV-Ab test during screening with positive HCV-RNA).
10. Other conditions considered by the investigator to potentially affect patient compliance or make the patient unsuitable for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Tumor assessments performed at baseline, then every 6-12 weeks from the start of treatment until disease progression or study completion (up to 24 months).
  The proportion of participants achieving a complete response (CR) or partial response (PR) based on modified RECIST v1.1 (mRECIST) criteria for target lesions assessed via MRI or CT imaging.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From the start of treatment until the first documented progression or death from any cause (assessed up to 24 months).
  The time from the start of treatment to the first occurrence of disease progression as per mRECIST criteria or death from any cause, whichever occurs first.
Overall Survival (OS) | From the start of treatment until death from any cause (assessed up to 24 months).
  The time from the start of treatment to death from any cause.
Incidence of Treatment-Related Adverse Events (AEs) | From the first administration of H101/TACE until 60 days after the last administration.
  The frequency and severity of adverse events assessed according to CTCAE v5.0, including those related to the oncolytic virus H101 and transarterial chemoembolization (TACE), such as injection site reactions, flu-like symptoms, myelosuppression, and procedural complications.

OTHER OUTCOMES:
Change in Quality of Life (QoL) Score | Assessed at baseline, then every 4-8 weeks from the start of treatment until disease progression or study completion (up to 24 months).
  The change from baseline in the Global Health Status / Quality of Life scale (Items 29 & 30) of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30. This scale consists of two items rated on a 7-point Likert scale (1='Very poor' to 7='Excellent'). The raw score is linearly transformed to a 0 to 100 scale, with a higher score indicating a better quality of life.
Change in Head and Neck Cancer-Specific Symptoms | Assessed at baseline, then every 4-8 weeks from the start of treatment until disease progression or study completion (up to 24 months).
  The change from baseline in the total symptom score of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck Cancer Module 35. The QLQ-H&N35 assesses symptoms and side effects specific to head and neck cancer and its treatment across multiple domains. Items are rated on a 4-point Likert scale (1='Not at all' to 4='Very much'). Scores are linearly transformed to a 0 to 100 scale, with a higher score indicating more severe symptoms or problems.